CLINICAL TRIAL: NCT02360371
Title: A118G SNP and OPRM1 Gene Opioid-Mediated Effects in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00047423; R01DA035246-01A1 (NIH)
Record Dates: First submitted 2015-01-29; First posted 2015-02-10 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Opioid Sensitivity; Individual Difference; Abuse Opioids
Keywords: opioid; abuse; genetic; A118G; OPRM1
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Within-subject, double-blind, randomized, placebo-controlled, human laboratory design wherein each participant completed each of the study conditions (outlined below as four arms). Participants were genotyped for rs-1799971and data were analyzed using between-group designs based upon rs-1799971 status.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants nor staff were informed of the class of drugs under investigation. Strict blinding was maintained.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (oral) (Placebo Comparator): Within-subject double-blind, administration of placebo oral capsule. Order of dose randomized session days 3-5.
  Interventions: Drug: Within-subject test of blinded study medication
- Hydromorphone (oral) 2mg (Experimental): Within-subject double-blind, administration of hydromorphone via oral capsule. Order of dose randomized session days 3-5.
  Interventions: Drug: Within-subject test of blinded study medication
- Hydromorphone (oral) 4mg (Experimental): Hydromorphone oral capsule administered in double-blind manner on Day 2 as first study drug administration. Hydromorphone 4mg dosing day was set for safety purposes and non-randomized.
  Interventions: Drug: Within-subject test of blinded study medication
- Hydromorphone (oral) 8mg (Experimental): Within-subject double-blind, administration of hydromorphone via oral capsule. Order of dose randomized session days 3-5.
  Interventions: Drug: Within-subject test of blinded study medication

INTERVENTIONS:
Drug: Within-subject test of blinded study medication — Within-subject double-blind, randomized, placebo-controlled, residential human abuse potential study. All participants received 4mg oral hydromorphone on study day 2 and a subset continued into the randomized portion for study days 3-5 wherein they received placebo, 2mg hydromorphone, and 8mg hydromorphone in randomized order. Only one dose was administered per day and following randomized all participants received each dose in random order. Outcomes were collected during 8-hour residential-based sessions and included metrics of FDA human abuse potential testing as well as secondary outcomes of laboratory pain testing, subjective reports of drug effects, and cognitive performance, evaluated as a function of study medication condition. Participants were genotyped for rs-1799971 status and results were analyzed as between-group comparisons based upon genotype.

SUMMARY:
Within-subject, double-blind, placebo-controlled examination of opioid abuse potential in healthy individuals as a function of A118G SNP on the OPRM1 gene.

DETAILED DESCRIPTION:
Participants completed a 5-day, within-subject, double-blind, placebo-controlled, randomized, human laboratory abuse potential trial. Healthy individuals were admitted to a residential research unit for 5 consecutive days. Blood samples were drawn for genome wide analyses using the Global Screening Array on day 1. Participants were administered an oral dose of the opioid hydromorphone (4mg) on day 2 of the study. Persons who did not evidence strong agonist effects then proceeded into the randomized period wherein they received 0mg, 2mg, and 8mg of oral hydromorphone on the remaining three study days. The order of dosing was randomized, with only 1 dose administered per day and all participants receiving 1 exposure to each dose. Outcomes were standard human abuse potential metrics, including self-reported drug effects and feeling high. Data were analyzed as a function of the A118SNP on the OPRM1 gene that codes for the mu opioid receptor. The overall aim was to determine whether signal for abuse potential among persons with no history of opioid misuse was associated with genotype.

ELIGIBILITY:
Inclusion Criterion:

1. Provide a urine sample that tests negative for opioids, methadone, buprenorphine, oxycodone, amphetamine, cocaine, and benzodiazepines
2. Negative ethanol breath test (0.000)
3. Aged 21-50
4. Deemed medically eligible to take hydromorphone

Exclusion Criterion:

1. Answer "yes" to question 1 of the Brief Pain Inventory (89) to assess the presence of chronic pain.
2. Current use of opioids or other medications for pain
3. Meet DSM-5 criteria for current or lifetime alcohol or drug use disorder (excluding nicotine)
4. Self-report any illicit drug use in the past 7 days
5. Self-report opioid use >5 days in the past 30
6. Evidence of opioid physical dependence at screening or following 1st residential overnight (following confirmed opioid abstinence)
7. Allergy to hydromorphone or other opioid agonists
8. Experience an adverse event that warrants opioid antagonist treatment following 1st hydromorphone dose.
9. If female, not be pregnant or breastfeeding
10. Presence of any clinically significant medical (e.g., chronic renal insufficiency, history of myocardial infarction, seizure disorder) and/or psychiatric illness (e.g., schizophrenia, bipolar disorder) that may interfere with study participation.
11. BMI >30 (obese category)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Dunn, Ph.D., MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Bayview Medical Campus, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Dunn KE, Huhn AS, Finan PH, Mange A, Bergeria CL, Maher BS, Rabinowitz JA, Strain EC, Antoine D. Polymorphisms in the A118G SNP of the OPRM1 gene produce different experiences of opioids: A human laboratory phenotype-genotype assessment. Addict Biol. 2024 Jan;29(1):e13355. doi: 10.1111/adb.13355. PMID 38221808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 participants were recruited from the community for participation. Analyses were based upon OPRM1 rs-1799971 allele status (A, G), which was available for 97 participants. All participants completed the same 4 study arms.
Groups:
- A118G (rs1799971-G); A118A (rs1799971-A): This is a within-subject study wherein the same participants moved from one treatment arm to the next and results were analyzed posthoc as a function of genotype.
Period: Overall Study
Arm/Group | A118G (rs1799971-G) | A118A (rs1799971-A)
Started | 13 | 84
Placebo (Oral) | 13 | 69
Hydromorphone (Oral) 2mg | 13 | 69
Hydromorphone (Oral) 4mg | 13 | 69
Hydromorphone (Oral) 8mg | 13 | 69
Completed | 13 | 69
Not Completed | 0 | 15

BASELINE CHARACTERISTICS:
Groups:
- A118G (rs1799971-G); A118A (rs1799971-A): This is a within-subject study wherein the same 100 participants moved from one treatment arm to the next.
- Total: Total of all reporting groups
Arm/Group | A118G (rs1799971-G) | A118A (rs1799971-A) | Total
Number analyzed (Participants) | 13 | 84 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (10.0) | 33.3 (8.9) | 33.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 45 | 49
  Male | 9 | 39 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 10 | 79 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 2 | 43 | 45
  White | 9 | 28 | 37
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 84 | 97

OUTCOME MEASURES:

1. Primary Outcome: Self-report Visual Analog Ratings of HIGH
Description: Peak visual analog rating scale values of HIGH (rated on 0-100 scale with higher scores indicating higher feeling of being HIGH) collected at 30 minute intervals post-drug administration for 6 hours.
Time Frame: 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A118G (rs1799971-G) | A118A (rs1799971-A)
Number analyzed (Participants) | 13 | 84
score on a scale
  Placebo (oral) | 7.2 (13.2) | 6.6 (16.3)
  Hydromorphone (oral) 2mg | 4.5 (5.9) | 5.6 (15.4)
  Hydromorphone (oral) 4mg | 12.5 (19.8) | 18.4 (26.4)
  Hydromorphone (oral) 8mg | 25.5 (29.7) | 22.5 (27.2)
Statistical Analysis 1: Comparison: A118G (rs1799971-G) vs A118A (rs1799971-A); Test type: Superiority; p = 0.567, Mixed methods

2. Primary Outcome: Self-report Visual Analog Ratings of DRUG EFFECT
Description: Peak visual analog rating scale values of DRUG EFFECT (rated on 0-100 scale with higher scores indicating higher drug effect) collected at 30 minute intervals post-drug administration for 6 hours.
Time Frame: 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A118G (rs1799971-G) | A118A (rs1799971-A)
Number analyzed (Participants) | 13 | 84
score on a scale
  Placebo (oral) | 13.3 (21.3) | 11.1 (20.0)
  Hydromorphone (oral) 2mg | 10.8 (16.5) | 11.0 (20.7)
  Hydromorphone (oral) 4mg | 23.6 (27.0) | 31.9 (29.9)
  Hydromorphone (oral) 8mg | 39.2 (37.3) | 39.5 (32.1)
Statistical Analysis 1: Comparison: A118G (rs1799971-G) vs A118A (rs1799971-A); Test type: Superiority; p = 0.805, Mixed Model

ADVERSE EVENTS:
Time Frame: Adverse events collected for 6 hours post each drug administration session. Only adverse events (AEs) judged to be possibly, probably, or definitely related to study participation are reported.
Description: AEs were documented the end of each session or in response to spontaneous reporting from participants, as a function of dose but not allele status, during the session. AEs were queried by asking "are you experiencing any side effects of the study medication?" The 4mg hydromorphone dose was the safety test dose and all individuals who had strong agonist responses (e.g., vomiting) in response to that dose were discontinued; therefore more individuals received 4mg than did other doses.
Arm/Group | Placebo (Oral) | Hydromorphone (Oral) 2mg | Hydromorphone (Oral) 4mg | Hydromorphone (Oral) 8mg
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82 | 0/97 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 0/97 | 0/82
Other Adverse Events (participants affected / at risk) | 19/82 | 21/82 | 65/97 | 49/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Oral) (N=82) | Hydromorphone (Oral) 2mg (N=82) | Hydromorphone (Oral) 4mg (N=97) | Hydromorphone (Oral) 8mg (N=82)
Headache (General disorders) | 5 (5) | 8 (8) | 6 (6) | 6 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 14 (16) | 7 (8)
Dry Mouth (Xerostomia) (General disorders) | 1 (1) | 0 (0) | 5 (6) | 6 (6)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 8 (11) | 9 (10)
Drowsiness (Nervous system disorders) | 10 (17) | 10 (13) | 31 (48) | 20 (35)
Euphoria/High (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Fatigue (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Impaired, Groggy (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Lethargy (Nervous system disorders) | 2 (4) | 1 (1) | 9 (10) | 1 (2)
Light Headedness (Nervous system disorders) | 1 (1) | 1 (1) | 10 (12) | 7 (7)
Shaky (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (3)
Sleepiness (Nervous system disorders) | 1 (1) | 2 (2) | 8 (9) | 4 (4)
Sluggish (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Pruritus (Itching) (Nervous system disorders) | 0 (0) | 2 (2) | 4 (5) | 8 (10)
Hot Flashes (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 29 (39) | 18 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT02360371/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT02360371/ICF_001.pdf